CLINICAL TRIAL: NCT05090540
Title: Transcatheter Edge to Edge Mitral Valve Repair Versus Standard Surgical Mitral Valve Operation for Secondadry Mitral Regurgitation
Brief Title: Transcatheter Versus Standard Surgical Mitral Valve Operation for Secondary Mitral Regurgitation
Acronym: TEERMISO
Status: Enrolling by invitation | Type: Observational
Sponsor: Centre Cardiologique du Nord (Other)
Collaborators: Campus Bio-Medico University (Other); Henri Mondor University Hospital (Other); Hokkaido University (Other); University of Genova (Other)
Responsible Party: Principal Investigator, Francesco Nappi, Principal Investigator, Centre Cardiologique du Nord
Other Study IDs: CN-21-23; CN-21-23 (Registry Identifier: TEERMISO)
Record Dates: First submitted 2021-09-23; First posted 2021-10-22 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Severe Mitral Valve Regurgitation (Disorder)
Keywords: SMR; TEER; MVRpl; MVR; RMA; Subvalvular Repair
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Transcatheter Edge to Edge Repair: TEER procedure is performed by apposing the edges of the anterior and posterior leaflet (edge-to-edge) of MV. If the use of one MitraClip device does not result in sufficient reduction in mitral regurgitation, a second MitraClip device may be used to reduce MR optimizing the procedure.
  Interventions: Device: Trancatheter Edge to Edge Repair
- Mitral Valve Replacement: Mitral-valve replacement includes complete preservation of the subvalvular apparatus to avoid dilation of the left ventricle over time. The technique of preservation, type of prosthetic valve implanted, and technique of suture placement has been chosen according to the preference of the surgeons. In SMR due to ischemic cardiomyopathy, CABG operation(Revascularization) is required
  Interventions: Procedure: Mitral Valve Replacement
- Restrictive Mitral Annuloplasty: RMA may be performed with the use of complete rigid or semi-rigid annuloplasty ring which has been downsized for the annulus diameter. Since patients who received RMA have coronary artery lesions, a CABG operation is useful to ensure favorable remodeling of the left ventricle.
  Interventions: Procedure: Restrictive Mitral Annuloplastie
- Restrictive Mitral Annuloplastie Plus Subvalvular Repair: RMA may be associated with the use of a subvalvular repair (SVR). The SVR permits the approximation or the relocation of papillary muscles which is displaced by post infarction scar formation. In patients who received SVR due to ischemic cardiomyopathy CABG operation is required
  Interventions: Procedure: Restrictive Mitral Annuloplastie/Subvalvular Repair

INTERVENTIONS:
Device: Trancatheter Edge to Edge Repair — TEER is performed by apposing the edges of the anterior and posterior leaflet (edge-to-edge) of prolapsed MV. The patient may be under conscious sedation or general anesthesia, depending on hospital standard practice. The procedure is performed through femoral venous access and the inter-atrial septum is crossed using standard techniques. Trans-septal puncture allows MitraClip Steerable Guide Catheter (Guide) to advance so that the guide is positioned over the mitral valve. The MitraClip delivery catheter is advanced to the MitraClip device and emerges from the tip of the guide into the left atrium. The MitraClip device can now be opened and advanced through the MV in the LV. Once in the LV, it is pulled back to grasp the leaflets. Two-dimensional and/or 3-dimensional echocardiography and color Doppler are useful for evaluating the anatomical features of the mitral valve and directing the procedure until the double orifice is formed alongside evaluating residual mitral regurgitation
  Other Names: Mitraclip procedure
  Groups: Transcatheter Edge to Edge Repair
Procedure: Mitral Valve Replacement — Mitral valve replacement is performed using mechanical or biological prosthesis while preserving the subvalvular apparatus to avoid dilation of the left ventricle over time.
  Groups: Mitral Valve Replacement
Procedure: Restrictive Mitral Annuloplastie — Mitral valve repair consists of a restrictive mitral annuloplasty (RMA) using a prosthetic ring
  Other Names: Undersizing Mitral Annuloplastie
  Groups: Restrictive Mitral Annuloplasty
Procedure: Restrictive Mitral Annuloplastie/Subvalvular Repair — RMA may be associated with the use of a subvalvular repair (SR). The SR permits the approximation or the relocation of papillary muscles which is displaced by post infarction scar formation.
  Groups: Restrictive Mitral Annuloplastie Plus Subvalvular Repair

SUMMARY:
The mechanical intervention is treating secondary mitral regurgitation (SMR) which may be performed using the standard open surgical approach or transcatheter edge to edge repair (TEER). The key question of this study is to establish the difference in left ventricular reverse remodeling after adjustment for death, as assessed by means of the left ventricular end-systolic dimension(LVESD), all-cause and cause-specific (cardiac vs noncardiac) mortality in patients who received the TEER vs the standard surgical procedure for SMR.

DETAILED DESCRIPTION:
The target population enrolled in the registry includes patients with moderate to severe secondary mitral regurgitation due to cardiomyopathy of either ischemic or non-ischemic etiology who have had TEER or standard surgical procedure of their mitral valves with or without CABG. Individuals were adequately treated per applicable standards, including for coronary artery disease, LV dysfunction, mitral regurgitation, and heart failure. Patients enrolled in the studies were NYHA functional class II, III, or outpatient NYHA IV.

Four groups of patients are included in the study. Patients who were managed with TEER, patients who received mitral valve replacement and recipients of mitral valve repair who underwent surgery with the use of restrictive annuloplasty alone or combined with subvalvular repair. Four groups of patients are included in the study. Patients who were managed with TEER, patients who received mitral valve replacement, and those who received mitral valve repair who underwent surgery with the use of restrictive annuloplasty alone or combined with subvalvular repair

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Ischemic NoIschemic cardiomyopathy
* EROA> 0,2 cm2 or Regurgitant Volume > 30 ml (ESC guidelines).
* EROA ≥ 0.4 cm2 with tethering (ACC/AHA)
* MR Grade 3/4
* Eligible for TEE, surgical repair and replacement of mitral valve
* Coronary artery disease with or without the need for coronary revascularization
* Average value LVEDD 62 mm LVEF 42%

Exclusion Criteria:

* Pediatric
* Any echocardiographic evidence of structural (chordal or leaflet) mitral-valve disease
* ruptured papillary

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with severe secondary mitral regurgitation with or without multivessel coronary artery disease who were symptomatic for congestive heart failure and unresponsive to medical therapy were eligible for surgical repair or replacement combined or not to coronary artery bypass graft (CABG). The severity of SMR was evaluated by transthoracic echocardiography, which was performed using European Society of Echocardiography criteria. Severe MR was defined as an effective regurgitant orifice area (EROA) of at least 0.4 cm2 or by a combination of adjunctive echocardiographic quantification methods according to guidelines. MR grade was defined according to EROA.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular Reverse Remodelling | 5 years
  The primary end point of the study is the degree of left ventricular reverse remodeling, as assessed by means of the left ventricular end systolic dimension on the basis of transthoracic echocardiography

SECONDARY OUTCOMES:
Overall Mortality | 5 years
  The secondary endpoint of the study is the evaluation of overall mortality
Cardiac Death | 5 years
  The secondary endpoint of the study is the evaluation of cardiac death
Major Adverse Cardiac or Cerebrovascular Events (MACCE) | 5 years
  Composite of major adverse cardiac or cerebrovascular events (rate of death, stroke, subsequent mitral valve surgery, hospitalization for heart failure, or an increase in New York Heart Association class higher than one), serious adverse events, recurrent mitral regurgitation, quality of life, and rehospitalization.
Echocardiographic Parameter Changes (LVEF) | 5 years
  Changes from baseline parameters including left ventricular ejection fraction
Echocardiographic Parameter Changes (recurrence) | 5 years
  Recurrent moderate-to-severe mitral regurgitation after intervention
Echocardiographic Parameter Changes (LVEDD) | 5 years
  Changes from baseline Left Ventricular End Diastolic Diameter
Echocardiographic Parameter Changes (Mitral Valve tenting area and height) | 5 years
  Changes from baseline tenting area and height
Echocardiographic Parameter Changes (Pulmonary artery systolic pressure) | 5 years
  Changes from baseline pulmonary artery systolic pressure
Echocardiographic Parameter Changes (anteroposterior mitral valve annular diameter) | 5 years
  Changes from baseline anteroposterior mitral valve annular diameter
Echocardiographic Parameter Changes ( interpapillary distance) | 5 years
  Changes from baseline distance between papillary muscles

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Nappi, MD, Principal Investigator — Centre Cardiologique du Nord
Locations (2):
- France (2):
  - Francesco Nappi, Saint-Denis
  - Centre Cardiologique Du Nord, Saint-Denis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nappi F, Singh SSA, Salsano A, Spadaccio C, Shingu Y, Wakasa S, Fiore A. Study protocol for an international registry observational study evaluating clinical outcomes of transcatheter versus standard surgical mitral valve operation for secondary mitral regurgitation: the TEERMISO study. BMJ Open. 2025 Jan 8;15(1):e086888. doi: 10.1136/bmjopen-2024-086888. PMID 39779262
- [Derived] Nappi F, Avtaar Singh SS, Salsano A, Nassif A, Shingu Y, Wakasa S, Fiore A, Spadaccio C, El-Dean Z. A Protocol Investigation Comparing Transcatheter Repair with the Standard Surgical Procedure for Secondary Mitral Regurgitation. J Clin Med. 2024 Dec 18;13(24):7742. doi: 10.3390/jcm13247742. PMID 39768667